CLINICAL TRIAL: NCT05603871
Title: The Role of Ligamentoplasty of Ligamentum Tere in the Management of Developmental Dysplasia of the Hip
Brief Title: Ligamentoplasty of Ligamentum Tere Developmental Dysplasia of the Hip
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Obeid Abd Allah, Principal Investigator, Al-Azhar University
Other Study IDs: LPLT
Record Dates: First submitted 2022-10-29; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ligamentoplasty of ligamentum teres: The patients will be examined for:
  1. Length of both lower limbs in relation to each other.
  2. Length of both lower limbs according to patient age.
  3. Presence of hump related to the outer surface of the hip
  4. Presence of pain, abnormal gait, Trendlenburg test.
  An addition to the steps of the open reduction, the following were done:
  1. Identification of ligamentum teres
  2. Ligamentoplasty of ligamentum teres
  Interventions: Procedure: ligamentoplasty of ligamentum teres

INTERVENTIONS:
Procedure: ligamentoplasty of ligamentum teres — An addition to the steps of the open reduction, the following were done:
  1. Identification of ligamentum teres
  2. Ligamentoplasty of ligamentum teres

SUMMARY:
The hip is formed by the acetabulum, the proximal femur and soft tissues joining them (capsule, teres ligament, transverse ligament and pulvinar). The acetabulum is a complex structure in the growing child. It is formed by the joined pubis, This junction is called tri radiate cartilage, which is responsible for acetabular growth. The external surface of the acetabulum is covered by a horse shoe-shaped articular cartilage. The transverse ligament joins both extremes of the articular cartilage inferiorly.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Developmental dysplasia of the hip (DDH) with :

  * Age: from 9 months -3 years old.
  * Virgin DDH.
  * Failed closed reduction in the management of DDH.
  * Failed open reduction through medial approach in the management of DDH.

Exclusion Criteria:

* • Paralytic hip dislocation .

  * Post septic hip dislocation.
  * Traumatic hip dislocation .
  * Age : below 9 months or above 5 years.
  * Refusal to participate in this study.

Ages: 9 Months to 3 Years | Sex: All
Age Groups: Child
Study Population: The patients will be examined for:
  Length of both lower limbs in relation to each other. Length of both lower limbs according to patient age. Presence of hump related to the outer surface of the hip Presence of pain, abnormal gait, Trendlenburg test Radiographic evaluation (antero posterior and frog pelvis views)
  An addition to the steps of the open reduction, the following were done:
  Identification of ligamentum teres and ligamentoplasty
Sampling Method: Non-Probability Sample
Enrollment: 3 (Estimated)
Dates: Start 2022-11-29 (Estimated); Primary Completion 2023-11-29 (Estimated); Study Completion 2023-11-29 (Estimated)

PRIMARY OUTCOMES:
modified Harris Hip Score | 6 months
  score for function of the hip

REFERENCES:
- [Background] Zhang S, Doudoulakis KJ, Khurwal A, Sarraf KM. Developmental dysplasia of the hip. Br J Hosp Med (Lond). 2020 Jul 2;81(7):1-8. doi: 10.12968/hmed.2020.0223. Epub 2020 Jul 6. PMID 32730146
- [Background] Schaeffer EK, Study Group I, Mulpuri K. Developmental dysplasia of the hip: addressing evidence gaps with a multicentre prospective international study. Med J Aust. 2018 May 7;208(8):359-364. doi: 10.5694/mja18.00154. PMID 29716513